CLINICAL TRIAL: NCT05260697
Title: The Effect of Sexual Counseling Based on PLISSIT Model to Women Undergoing Open Heart Surgery on Sexual Function and Sexual Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Merve Tuncer, Lecturer, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 13022260-302.14.05
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: PLISSIT Model; Sexual Counselling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sexual Counselling Group (Experimental): Sexual Counselling with PLISSIT model
  Interventions: Other: sexual counselling with plissit model
- Control Group (No Intervention): no intervention group

INTERVENTIONS:
Other: sexual counselling with plissit model — sexual counselling
  Arms: Sexual Counselling Group

SUMMARY:
This study is about sexual counseling after cardiac surgery; It can contribute to the counseling planning of nurses and other health professionals regarding sexual problems that may occur after surgery. Increasing the quality of life in the rehabilitation process after cardiac surgery and facilitating adaptation to life after surgery; but not enough.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Being a woman
* Being over 18 years old
* Willingness to undergo open heart surgery
* Euroscore score ≤ 6 (low mortality risk due to cardiac surgery)
* Being sexually active
* Absence of sexual health problems in the spouse
* Ability to communicate verbally and be literate
* Women without neurological or psychiatric disorders
* Knowing Turkish

Exclusion Criteria:

* Unwillingness to participate in the research
* Euroscore score >6 (high risk of mortality)
* Not being sexually active
* Having a diagnosed sexual health problem in the spouse
* Women with neurological and psychiatric disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women gender
Enrollment: 64 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
'Female Sexual Function Index' scores will increase after sexual counseling based on the PLISSIT model will be given to individuals who will undergo open heart surgery. | 1 year
After the sexual counseling based on the PLISSIT model to be given to the individuals who will undergo open heart surgery, the scores of the "Sexual Quality of Life Scale-Female Form" will increase. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Merve TUNCER, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tuncer M, Yesiltepe Oskay U. Effect of sexual counseling on sexual function and sexual quality of life for women undergoing open heart surgery: a pilot randomized controlled trial. J Sex Med. 2023 Jun 28;20(7):1010-1017. doi: 10.1093/jsxmed/qdad065. PMID 37246308